CLINICAL TRIAL: NCT07015138
Title: A Multicenter, Randomized Controlled Clinical Trial Comparing Comprehensive Radiotherapy Versus Primary Tumor Radiotherapy in Oligometastatic Prostate Cancer
Brief Title: Comprehensive Versus Primary Tumor Radiotherapy in Oligometastatic Prostate Cancer
Acronym: PROLONG-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROLONG-3
Record Dates: First submitted 2025-05-20; First posted 2025-06-11 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer; Oligometastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study established a blinded assessment and endpoint adjudication committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A (Experimental): Comprehensive Radiotherapy + Standard Systemic Therapy
  Interventions: Radiation: TRT
- Arm B (Active Comparator): Primary Radiotherapy + Standard Systemic Therapy
  Interventions: Radiation: NTRT

INTERVENTIONS:
Radiation: TRT — Comprehensive metastasis-directed radiotherapy:
  * Targets: Primary prostate tumor + all metastatic lesions (≤10 sites confirmed by PSMA PET)
  * Concurrent therapy: Standard systemic treatment (ADT + novel hormonal agents)
  Arms: ARM A
Radiation: NTRT — Standard primary radiotherapy:
  * Targets: Prostate primary tumor only
  * Concurrent therapy: Same systemic treatment as experimental arm
  Arms: Arm B

SUMMARY:
This study is a multicenter, randomized controlled phase III clinical trial (PROLONG-3) designed to evaluate the survival benefit of comprehensive radiotherapy combined with primary tumor radiotherapy versus primary tumor radiotherapy alone in patients with newly diagnosed oligometastatic prostate cancer. The trial enrolled 390 patients with ≤10 metastatic lesions confirmed by PSMA PET imaging, who were randomized in a 2:1 ratio to either the intervention group (comprehensive radiotherapy + standard systemic therapy) or control group (primary radiotherapy + standard systemic therapy).

Stratification factors included Gleason score (GS ≤8 vs. GS 9-10) and number of metastases (1-3 vs. 4-10). The primary endpoint was 3-year progression-free survival (PFS), with secondary endpoints encompassing overall survival (OS), intermittent treatment rate, adverse events (CTCAE v5.0), and quality of life (EORTC QLQ questionnaires). To minimize bias, stratified block randomization and blinded endpoint adjudication were implemented, with treatment effects analyzed using Kaplan-Meier survival curves and Cox proportional hazards models.

The study's innovation lies in its definitive evaluation of the added value of comprehensive radiotherapy, combined with exploratory biomarker analyses (including genomic testing) to identify predictive markers of therapeutic response. Should the results demonstrate significant PFS improvement with comprehensive radiotherapy, this would provide high-level evidence to guide clinical practice, potentially influencing treatment guideline updates while optimizing patient quality of life and reducing healthcare burdens.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18-85 years.
* Histopathologically confirmed acinar adenocarcinoma of the prostate. The presence of a minor component of ductal adenocarcinoma, intraductal carcinoma, and/or neuroendocrine differentiation is permitted.
* PSMA PET performed within 4 weeks prior to the start of study drug therapy or up to 4 weeks after initiation, demonstrating the presence of 1 to 10 metastatic lesions.Metastasis within pelvic lymph nodes (N1 disease) is permitted but not counted towards the total number of metastatic lesions. Metastasis to non-regional lymph nodes is permitted and counted towards the total number.The pelvis is anatomically divided into 4 regions: left hemipelvis (ilium/ischium/pubis), right hemipelvis (ilium/ischium/pubis), sacrum, and coccyx. Multiple lesions within a single anatomical division are aggregated and counted as one metastatic lesion.
* Prior androgen deprivation therapy (ADT) is permitted if the total duration was ≤ 12 months before enrollment. ADT includes luteinizing hormone-releasing hormone (LHRH) agonists or antagonists and novel hormonal agents (e.g., abiraterone, enzalutamide, apalutamide, darolutamide).
* Eastern Cooperative Oncology Group (ECOG) score 0-2.
* Hematology: Neutrophil count >=1.0×10^9/L; Platelet count >=75×10^9/L; Hemoglobin >=90 g/L.

Exclusion Criteria:

* Small cell carcinoma of the prostate or prostate sarcoma.
* The primary focus has received external radiation therapy, brachytherapy, and radical prostatectomy.
* Received non-endocrine systemic therapies prior to enrollment (e.g., chemotherapy, targeted therapy, radionuclide therapy).
* Metastatic castration-resistant prostate cancer (mCRPC) phase (EAU Guidelines*).
* Presence of visceral metastases (e.g., liver, lung).
* Previous bilateral orchiectomy.
* Comorbidities: Severe comorbidities affecting survival or treatment tolerance, including: Cardiovascular diseases (NYHA Class III/IV heart failure, uncontrolled arrhythmias); Renal insufficiency (eGFR <30 mL/min/1.73m^2); Neuropsychiatric disorders impairing protocol compliance.

  * Definition of mCRPC (EAU Guidelines):

Metastatic castration-resistant prostate cancer (mCRPC) is defined as disease progression despite serum testosterone levels below 50 ng/dL (or 1.7 nmol/L), concurrently with one or more of the following:

1. PSA progression: A sequence of at least three consecutive rises in PSA, measured ≥1 week apart, resulting in a ≥50% increase from the nadir (lowest) level, with a minimum absolute PSA value >2 ng/mL.
2. Radiographic progression: The appearance of new lesions, defined as either:

   * ≥2 new lesions on bone scan (Tc-99m bone scintigraphy), or
   * New measurable soft tissue lesions according to RECIST (Response Evaluation Criteria in Solid Tumors) 1.1 criteria.
3. Unequivocal clinical progression: Clinical progression in the absence of concurrent PSA or radiographic progression should be viewed with suspicion and mandates further investigation to confirm disease progression.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year progression-free survival (PFS) | Post-radiotherapy follow-up at 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, and 36 months

SECONDARY OUTCOMES:
Time to PSA progression | Post-radiotherapy follow-up at 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, and 36 months
Overall survival (OS) | Post-radiotherapy follow-up at 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, and 36 months
3-year treatment discontinuation rate | Post-radiotherapy follow-up at 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, and 36 months
Quality of life (QoL) | Post-radiotherapy follow-up at 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, and 36 months
  Measure Tools:
  EORTC QLQ-C30 (Version 3.0): Global health status (Items 29-30), functional scales (physical, role, emotional, cognitive, social), and symptom scales (fatigue, pain, nausea, etc.).
  Scale Range: 0-100 for all domains. Interpretation: Higher scores = better functioning (global/functional scales) or worse symptoms (symptom scales).
  QLQ-PR25: Prostate cancer-specific module (symptoms, treatment side effects, sexual function).
  Scale Range: 0-100 for all subscales
  Interpretation:
  Higher scores = worse symptoms (urinary, bowel, treatment-related). Sexual Activity Subscale: Higher scores = more sexual activity (better functioning).
  Sexual Functioning Subscale: Higher scores = worse sexual function (e.g., erectile dysfunction).
Adverse events (AEs) / Toxicity | Post-radiotherapy follow-up at 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, and 36 months
Time to initiation of subsequent anti-tumor therapy | Post-radiotherapy follow-up at 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, and 36 months
3-year treatment discontinuation rate (in patients with normalized testosterone) | Post-radiotherapy follow-up at 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, and 36 months
Radiographic progression-free survival (rPFS) | Post-radiotherapy follow-up at 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, and 36 months
Complete PSA response rate | 6 months after radiotherapy
  Definition: According to Prostate Cancer Working Group 3 (PCWG3) criteria, the following conditions must be met:
  PSA level decreases to undetectable levels (≤0.2 ng/mL). Confirmed by two consecutive measurements (≥4 weeks apart) with no clinical/radiographic progression (per RECIST 1.1).
  Measurement Tools:
  PSA Assay Method: Electrochemiluminescence immunoassay (ECLIA) or isotope dilution liquid chromatography-mass spectrometry (ID-LC/MS), with a lower limit of quantification (LLoQ) of 0.02 ng/mL.
  Radiographic Confirmation: Exclude disease progression (bone scan/CT/MRI per RECIST 1.1).
  Statistical Analysis:
  Proportion (%) of patients meeting the above criteria, with two-sided 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Hong-zhen Li, Study Chair — Peking University First Hospital
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No